CLINICAL TRIAL: NCT03337828
Title: Randomized, Cross-over Study Comparing the Effect of Two Alcohol-free Beers With Different Carbohydrates Composition on Lipid and Glycemic Metabolism in Subjects With Prediabetes and Recently Diagnosed Diabetes and Overweight or Obesity
Brief Title: Effect of Two Alcohol-free Beers With Different Carbohydrates Composition on Lipids and Glucose Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Aragon Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Fernando Civeira, Professor of Medicine, Aragon Institute of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEICA PI16/0277
Record Dates: First submitted 2017-10-31; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus); Overweight and Obesity
Keywords: Alcohol-free beer; Carbohydrates; Overweight; Obesity; Diabetes mellitus type 2; Microbiota; Glucose metabolism
MeSH Terms: conditions — Glucose Metabolism Disorders; Overweight; Obesity; Diabetes Mellitus, Type 2 | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol-free beer with regular composition (Active Comparator): Two cans (33 cl.) per day of an alcohol-free beer with regular carbohydrates composition.
  Interventions: Other: Alcohol-free beer with regular composition
- Alcohol-free beer with modified composition (Experimental): Two cans (33 cl.) per day of alcohol-free beer with modified carbohydrates composition. This include the substitution of regular maltose by isomaltulose and the addition of maltodextrin (fiber).
  Interventions: Other: Alcohol-free beer with modified composition

INTERVENTIONS:
Other: Alcohol-free beer with regular composition — Subjects are provided with 2 alcohol-free beers with regular carbohydrates composition per day and healthy diet counselling during 10 weeks.
  Arms: Alcohol-free beer with regular composition
Other: Alcohol-free beer with modified composition — Subjects are provided with 2 alcohol-free beers with modified carbohydrates composition per day and healthy diet counselling during 10 weeks.
  Arms: Alcohol-free beer with modified composition

SUMMARY:
This a controlled, double-blind, randomized, cross designed study to determine the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on glycemic metabolism (glucose, glycated hemoglobin, insulin and HOMA index) in subjects with recently diagnosed diabetes mellitus and overweight or obesity. 44 subjects were randomized to consume for 10 weeks: a) two alcohol-free beers with regular carbohydrates composition per day; b) two alcohol-free beers with modified carbohydrates composition per day. Those subjects randomized to begin with A beer during 10 weeks will change to B beer during the second phase for 10 weeks and vice versa. There is a 4-8 weeks wash-out period between two phases.

DETAILED DESCRIPTION:
The study involves a nutritional intervention with a controlled, double-blind, randomized, cross design. It includes 44 healthy subjects with a total duration of 20 weeks with a "wash-out/stabilization" period for 2-4 weeks before randomization. Subjects are randomized in two groups: (1) those who begin drinking 2 alcohol-free beers (33 cl each one) that are enriched in a resistant maltodextrin and isomaltulose during 10 weeks and continue drinking 2 alcohol-free beers (33 cl each one) with regular composition during the next 10 weeks following; (2) those who will follow the same previous intervention but in reverse, beginning with standard alcohol-free beer for 10 weeks, followed by resistant maltodextrin and isomaltulose-enriched beer for the remaining 10 weeks. There is a washout period between both phases to facilitate adherence to nutritional intervention, since we consider that a period of 20 consecutive weeks could be difficult to assume for the participants. Participants and the research team are "blind" to the type of beer that subjects are taking in each phase. Only one person of the company that provide beers, which does not directly participate in the clinic visits or in the analysis of the data, is aware of this information. Clinical staff performed the randomization based on a computerized method.

Among those subjects included in the study, microbiota sub-study is proposed which require a specific authorization within informed consent. Among all subjects that are included in this substudy and that have completed the whole nutritional intervention, 10 subjects (5 from each randomized group) will be selected to microbiota determination.

* Study visits:

  1. Prescreening visit: Inclusion and exclusion criteria assessment and blood collection if glucose or glycated hemoglobin is not available in previous 3 months. Healthy diet and physical activity counselling is provided by a nutritionist; it should be maintained during all study. Baseline visit is scheduled in 2-4 weeks after lifestyle stabilization.
  2. Baseline phase 1 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Computer-based randomization is performed. Alcohol-free beer (A or B according to randomization procedures) for the next 10 weeks is delivered to the participant who has to consume two per day. A nutritionist emphasizes healthy lifestyle counselling to the participant. A feces sample is collected if subjects accept to be included in microbiota sub study.
  3. Intermediate phase 1 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Satiety after alcohol-free beer consumption is measured by a validated questionnaire. A nutritionist emphasizes healthy lifestyle counselling to the participant.
  4. End of phase 1 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Satiety after alcohol-free beer consumption is measured by a validated questionnaire. A nutritionist emphasizes healthy lifestyle counselling to the participant. A wash-out period of 4-8 weeks is scheduled before the next phase start. A feces sample is collected if subjects accept to be included in microbiota sub study.
  5. Baseline phase 2 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Alcohol-free beer (A or B: if subjects consumed alcohol-free beer A, he/she change to alcohol-free B and vice versa) for the next 10 weeks is delivered to the participant who has to consume two per day. A nutritionist emphasizes healthy lifestyle counselling to the participant. A feces sample is collected if subjects accept to be included in microbiota sub study.
  6. Intermediate phase 2 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Satiety after alcohol-free beer consumption is measured by a validated questionnaire. A nutritionist emphasizes healthy lifestyle counselling to the participant.
  7. End of phase 2 visit: Clinical, biochemical, dietary, physical activity and anthropometric data are assessed. Satiety after alcohol-free beer consumption is measured by a validated questionnaire. A nutritionist emphasizes healthy lifestyle counselling to the participant. A feces sample is collected if subjects accept to be included in microbiota sub study.
* Study variables:

  * Clinical variables: Gender, age, medical records including diseases and medication, tobacco consumption and blood pressure.
  * Anthropometric variables: Weight, height, body mass index, waist circumference, body composition analysis.
  * Biochemical variables: Glucose, lipid and iron metabolism are assessed. Inflammatory biomarkers, including C reactive protein, are also determined.
  * Microbiota: Feces samples are collected to microbiota analysis including Bacteroides, Lactobacillus, Enterococcus, Prevotella or Roseburia, among others.
  * Dietary and physical activity assessment: Diet and physical activity are assessed by validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years.
* To provide informed consent in writing of voluntary participation in the study after having read the participant information sheet, and having consulted the doubts that may arise from it.
* Diagnosis of prediabetes or diabetes mellitus type 2 defined as: a) fasting glucose ≥ 100 mg/dL in the last 3 months; b) glycated hemoglobin ≥ 5.7% and ≤ 6.5%.

Exclusion Criteria:

* Gluten intolerance.
* Taking lipid-lowering drugs.
* Taking antidiabetic drugs, except for metformin in a stable dose in the last 3 months.
* To be under treatment with insulin.
* Presence of uncontrolled endocrinological disease by including hypothyroidism.
* Regular intake of functional foods with plant sterols in the past 6 weeks.
* Intake of vitamin supplements.
* Hormone replacement therapy.
* High intake of alcohol (> 30 g ethanol) on a regular basis.
* Pregnancy or intention of pregnancy during the study since the proposed nutritional intervention may not be suitable for this situation.
* Serious illness of any type with less than 1-year life expectancy or if, in the opinion of the investigators, it would limit a stable diet throughout the study.
* To be under treatment with corticosteroids, hormonal treatment or antibiotics the 3 months prior to randomization.
* To take prebiotics, probiotics, vitamin supplements and any other drug that could influence the intestinal microbiota, in the 3 months prior to randomization.
* Any other circumstances which, according to researcher's assessment, could interfere with the correct development of nutritional intervention (e.g.: frequent trips during the study, failure to attend visits by personal or business circumstances, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration change after each alcohol-free beer phase. | 10 weeks
  Main objective is to determine the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on glucose concentration change.
Glycated hemoglobin concentration change after each alcohol-free beer phase. | 10 weeks
  Main objective is to determine the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on glycated hemoglobin concentration change.
Insulin concentration change after each alcohol-free beer phase. | 10 weeks
  Main objective is to determine the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on insulin concentration change.
Homeostatic model assessment (HOMA) index change after each alcohol-free beer phase. | 10 weeks
  Main objective is to determine the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on HOMA index change.

SECONDARY OUTCOMES:
Lipid profile change after each alcohol-free beer phase. | 10 weeks
  Secondary objective involves determining the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on LDL cholesterol concentration change.
Body weight change after each alcohol-free beer phase. | 10 weeks
  Secondary objective involves determining the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on body weight.
C reactive protein concentration change after each alcohol-free beer phase. | 10 weeks
  Secondary objective involves determining the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on C reactive protein change.
Micriobota change after each alcohol-free beer phase. | 10 weeks
  Secondary objective involves determining the effect of an alcohol-free beer with low glycemic index carbohydrates (isomaltulose) and a resistant maltodextrin, comparing to an alcohol-free beer with regular composition, on microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Rocio Mateo-Gallego, RD, PhD, Principal Investigator — Aragon Institute of Health Sciences
Locations (1):
- Fernando Civeira, Zaragoza, Spain

REFERENCES:
- [Derived] Mateo-Gallego R , Moreno-Indias I , Bea AM , Sanchez-Alcoholado L , Fumanal AJ , Quesada-Molina M , Prieto-Martin A , Gutierrez-Repiso C , Civeira F , Tinahones FJ . An alcohol-free beer enriched with isomaltulose and a resistant dextrin modulates gut microbiome in subjects with type 2 diabetes mellitus and overweight or obesity: a pilot study. Food Funct. 2021 Apr 21;12(8):3635-3646. doi: 10.1039/d0fo03160g. Epub 2021 Mar 31. PMID 33900319
- [Derived] Mateo-Gallego R, Perez-Calahorra S, Lamiquiz-Moneo I, Marco-Benedi V, Bea AM, Fumanal AJ, Prieto-Martin A, Laclaustra M, Cenarro A, Civeira F. Effect of an alcohol-free beer enriched with isomaltulose and a resistant dextrin on insulin resistance in diabetic patients with overweight or obesity. Clin Nutr. 2020 Feb;39(2):475-483. doi: 10.1016/j.clnu.2019.02.025. Epub 2019 Mar 5. PMID 30879735

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT03337828/Prot_SAP_000.pdf